CLINICAL TRIAL: NCT01922271
Title: A Randomized, Double-blind, Multicenter, 2-period Single-dose Cross-over Study to Assess the Early Bronchodilation of Glycopyrronium Bromide (44 μg o.d.) Compared to Tiotropium (18 µg. o.d.) in Patients With Moderate to Severe COPD (FAST Study)
Brief Title: Efficacy of NVA237 Compared to Tiotropium in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Acronym: FAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNVA237ADE02
Record Dates: First submitted 2013-08-09; First posted 2013-08-14 (Estimated); Results first posted 2015-01-01 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate; Tiotropium Bromide; Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NVA237 followed by tiotropium (Experimental): Period 1: NVA237 plus placebo to tiotropium on day 1, followed by a 7 day washout. Period 2: tiotropium plus placebo to NVA237 on day 8. Salbutamol was used as rescue medication.
  Interventions: Drug: NVA237; Drug: Tiotropium; Drug: Placebo to tiotropium; Drug: Salbutamol
- Tiotropium followed by NVA237 (Experimental): Period 1: tiotropium plus placebo to NVA237 on day 1, followed by a 7 day washout. Period 2: NVA237 plus placebo to tiotropium on day 8. Salbutamol was used as rescue medication.
  Interventions: Drug: Placebo to NVA237; Drug: Salbutamol

INTERVENTIONS:
Drug: NVA237 — NVA237 44 µg inhalation capsules once daily, delivered via single-dose dry-powder inhaler (SDDPI)
  Arms: NVA237 followed by tiotropium
Drug: Tiotropium — Tiotropium 18 μg once daily delivered via HandiHaler® device.
  Arms: NVA237 followed by tiotropium
Drug: Placebo to NVA237 — Placebo to NVA237 once daily, delivered via single-dose dry-powder inhaler (SDDPI).
  Arms: Tiotropium followed by NVA237
Drug: Placebo to tiotropium — Placebo to tiotropium once daily delivered via HandiHaler® device
  Arms: NVA237 followed by tiotropium
Drug: Salbutamol — Used as resuce medication

SUMMARY:
The purpose of this study is to further figure out differences of glycopyrronium bromide compared to tiotropium in early bronchodilation measured by a comprehensive assessment of lung function that includes hyperinflation and specific airway resistance in patients with moderate to severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged ≥40 years
* Patients with moderate to severe COPD defined by a post-bronchodilator Forced Expiratory Volume in One Second (FEV1)/(FVC) Forced Vital Capacity ratio of <0.70 and a post-bronchodilator FEV1 of ≤70% and FEV1 ≥ 30% of predicted normal values.
* Current or ex-smokers who have a smoking history of at least 10 pack years.

Exclusion Criteria:

* Pregnant or nursing (lactating) women
* Patients who have a clinically significant laboratory abnormality at run-in
* Patients with narrow-angle glaucoma, symptomatic benign prostatic hyperplasia or bladder-neck obstruction or moderate to severe renal impairment (GFR <50 ml/min/1,732) or urinary retention. (BPH patients who are stable on treatment can be considered).
* Patients with any history of asthma
* Patients with pulmonary lobectomy or lung volume reduction surgery or lung transplantation
* Patients receiving medications in the classes listed in the protocol as prohibited.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2013-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- Germany (11):
  - Novartis Investigative Site, Leipzig, Germany
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Gelsenkirchen
  - Novartis Investigative Site, Großhansdorf
  - Novartis Investigative Site, Gummersbach
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Sonneberg

REFERENCES:
- [Derived] Watz H, Mailander C, May C, Baier M, Kirsten AM. Fast onset of action of glycopyrronium compared with tiotropium in patients with moderate to severe COPD - A randomised, multicentre, crossover trial. Pulm Pharmacol Ther. 2017 Feb;42:13-20. doi: 10.1016/j.pupt.2016.12.001. Epub 2016 Dec 9. PMID 27940287

RESULTS

PARTICIPANT FLOW:
Period: PERIOD 1
Arm/Group | NVA237 Followed by Tiotropium | Tiotropium Followed by NVA237
Started | 76 | 76
Completed | 76 | 76
Not Completed | 0 | 0
Period: WASHOUT Period
Arm/Group | NVA237 Followed by Tiotropium | Tiotropium Followed by NVA237
Started | 76 | 76
Completed | 75 | 76
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: PERIOD 2
Arm/Group | NVA237 Followed by Tiotropium | Tiotropium Followed by NVA237
Started | 75 | 76
Completed | 75 | 76
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NVA237 Followed by Tiotropium | Tiotropium Followed by NVA237 | Total
Number analyzed (Participants) | 76 | 76 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (7.2) | 61.7 (8.2) | 61.8 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 26 | 54
  Male | 48 | 50 | 98

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under Curve (AUC) 0-2
Description: Standardized Forced Expiratory Volume in One Second (FEV1) AUC0-2h will be measured via spirometry. The AUC will be calculated from the FEV1 measurements obtained at timepoints between 0 min and 2h using the trapezoidal rule and will be standardized (=divided) by the measurement time (i.e. 2h).
Time Frame: Day 1
Population: The Full Analysis Set (FAS) consisted of all randomized patients who applied at least one dose of study medication during at least one study period.
Measure: Mean (Standard Deviation); unit: liters per hour
Groups:
- NVA237: ALL patients on NVA237 for Period 1 & Period 2
- Tiotropium: ALL patients onTiotropium for Period 1 & Period 2
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 151 | 150
liters per hour | 1.490 (0.4232) | 1.453 (0.4135)

2. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) 15 Min Post Dose
Description: Forced expiratory volume in 1 second (FEV1) is the amount of air that can be exhaled in one second. FEV1 will be measured by spirometry. All spirometry calibrations and evaluations will follow the recommendations of the American Thoracic Society / European Respiratory Society guidelines for acceptability.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: liters per hour
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 152 | 151
liters per hour | 1.433 (0.4110) | 1.398 (0.4092)

3. Secondary Outcome: Specific Airway Resistance (sRAW)
Description: Specific Airway Resistance (sRAW) indicates volume and resistance-dependent work of breathing needed in order to generate a reference flow rate of 1 L/s, measured by kPa*s. Whole body plethysmography (Bodybox) is used to measure SRaw.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilopascal (kPa)
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 152 | 152
kilopascal (kPa)
  -45 min (n=152, 150) | 4.203 (1.8102) | 4.105 (1.8338)
  30 min (n=150, 151) | 2.904 (1.4759) | 3.089 (1.4555)
  1 hr (n=151, 149) | 2.656 (1.3062) | 2.877 (1.4130)
  1 hr 30 min (n=151, 150) | 2.632 (1.3152) | 2.811 (1.4065)
  2 hr 30 min (n=150, 149) | 2.643 (1.3146) | 2.756 (1.4091)
  3 hr 30 min (n=150, 149) | 2.779 (1.4496) | 2.828 (1.4534)

4. Secondary Outcome: Functional Resistance Capacity (FRCpleth)
Description: Functional Resistance Capacity (FRCpleth) will be measured using whole body plethysmography (Bodybox).
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 152 | 152
Liters
  -45 min (n=152, 150) | 5.211 (1.3086) | 5.142 (1.2656)
  30 min (n=150, 151) | 4.823 (1.2517) | 4.852 (1.1812)
  1 hr (n=151, 149) | 4.769 (1.2571) | 4.725 (1.1496)
  1 hr 30 min (n=151, 149) | 4.756 (1.2366) | 4.714 (1.1523)
  2 h 30 min (n= 150, 149) | 4.736 (1.1545) | 4.676 (1.2243)
  3 h 30 min (n= 150, 148) | 4.761 (1.2286) | 4.704 (1.1911)

5. Secondary Outcome: Residual Volume (RV)
Description: Residual Volume (RV) will be measured using whole body plethysmography (Bodybox).
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 152 | 152
Liters
  -45 min (n=152, 150) | 4.433 (1.2596) | 4.344 (1.1707)
  30 min (n=150, 151) | 3.996 (1.1862) | 4.035 (1.0689)
  1 hr (n=151, 149) | 3.891 (1.1997) | 3.913 (1.0281)
  1 hr 30 min (n=151, 149) | 3.910 (1.1534) | 3.903 (1.0281)
  2 h 30 min (n= 150, 149) | 3.893 (1.0486) | 3.861 (1.1058)
  3 h 30 min (n= 150, 148) | 3.970 (1.1576) | 3.895 (1.0740)

6. Secondary Outcome: Total Lung Capacity (TLC)
Description: Total Lung Capacity (TLC) is the best vital capacity plus residual volume (RV). Whole body plethysmography (Bodybox) will be used to measure TLC.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 152 | 152
Liters
  -45 min (n=152, 150) | 7.380 (1.4781) | 7.335 (1.4328)
  30 min (n=150, 151) | 7.255 (1.4628) | 7.274 (1.4032)
  1hr (n=151, 149) | 7.224 (1.4294) | 7.161 (1.4015)
  1hr 30 min (n=151, 149) | 7.227 (1.4383) | 7.165 (1.3690)
  2hr 30 min (n=150, 149) | 7.203 (1.3700) | 7.149 (1.4476)
  3hr 30 min (n=150, 148) | 7.240 (1.4297) | 7.149 (1.3963)

7. Secondary Outcome: Inspiratory Capacity (IC)
Description: Inspiratory Capacity (IC) is the volume of air breathed in by a maximum inspiration at the end of a normal expiration. Whole body plethysmography (Bodybox) will be used to measure IC.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | NVA237 | Tiotropium
Number analyzed (Participants) | 152 | 152
Liters
  -45 min (n=152, 150) | 2.169 (0.5548) | 2.193 (0.5583)
  30 min (n=150, 151) | 2.433 (0.5934) | 2.422 (0.5996)
  1hr (n=151, 149) | 2.455 (0.6001) | 2.435 (0.5908)
  1hr 30 min (n=151, 150) | 2.472 (0.6200) | 2.457 (0.5883)
  2hr 30 min (n=150, 149) | 2.467 (0.5929) | 2.474 (0.6051)
  3hr 30 min (n=150, 149) | 2.479 (0.6036) | 2.449 (0.5907)

ADVERSE EVENTS:
Arm/Group | NVA237 | Tiotropium
Serious Adverse Events (participants affected / at risk) | 2/152 | 2/151
Other Adverse Events (participants affected / at risk) | 8/152 | 15/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 (N=152) | Tiotropium (N=151)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nephrectomy (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 (N=152) | Tiotropium (N=151)
Condition aggravated (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 4
Rhinitis (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.